CLINICAL TRIAL: NCT00566930
Title: Preventive Care of Chronic Cervical Pain and Disabilities; Comparison of Spinal Manipulative Therapy and Individualized Home Exercise Programs
Brief Title: Preventive Care of Chronic Cervical Pain and Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Foundation for Chiropractic Education and Research (FCER) (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Chronic cervical pain UQTR; FCER Grant #06-03-02
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention)
- 2 (Active Comparator): spinal manipulation
  Interventions: Other: spinal manipulation
- 3 (Experimental): Spinal manipulation + exercises
  Interventions: Other: Spinal manipulation + exercises

INTERVENTIONS:
Other: spinal manipulation — Monthly cervical spinal manipulation
  Arms: 2
Other: Spinal manipulation + exercises — Monthly cervical spine manipulation and daily home exercises
  Arms: 3

SUMMARY:
The aim of this study is to determine which of tertiary prevention spinal manipulative therapy (SMT) or a home exercise program is the more efficient approach to reduce pain and increase functional capacity, quality of life and general health condition. To do so, 60 participants with chronic cervical pain, will be recruited and divided into 3 groups according to the intervention they will receive: control group, experimental group 1 who will receive preventive chiropractic care in the form of spinal manipulations and experimental group 2 will have to perform an individualized home exercise program on a daily basis. We hypothesize that a group of patient receiving SMT + a home exercise program will present less pain and functional disabilities over a 1 year period. The innovative value of this project is mainly related to the fact that it will generate new and potentially very useful data concerning the clinical significance of preventive chiropractic care. Moreover, such data will be beneficial to our profession as chiropractic makes a step towards prevention, wellness and public health.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 60 years old from the city and the surrounding Trois-Rivières with chronic cervical pain of non-traumatic origin (chronic or recurrent cervical pain that lasted at least 6 months)

Exclusion Criteria:

Exclusion criteria for the project are:

* Surgery to the cervical spine
* Neoplasms
* Severe osteoarthritis
* Ankylosing spondylitis
* Hypertension
* Referred pain in the cervical area
* Central or peripheric nervous system dysfunction
* Vascular disease
* Treated cardiovascular disease
* Inflammatory or infectious disease of the cervical spine
* Metabolic or endocrine diseases
* Pregnancy
* Specific rehabilitation training for the neck or already under manual therapy for neck pain
* Patient suffering from dizziness, vertigo or headache suspected to be cervicogenic or of unknown origin will not be involved in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Derived] Martel J, Dugas C, Dubois JD, Descarreaux M. A randomised controlled trial of preventive spinal manipulation with and without a home exercise program for patients with chronic neck pain. BMC Musculoskelet Disord. 2011 Feb 8;12:41. doi: 10.1186/1471-2474-12-41. PMID 21303529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: chripractic clinic
Pre-assignment Details: 117 participants were initially recruited. Following the initial clinical assessment, 98 met all inclusion criteria and were assigned to one of the three groups. 19 participants were excluded because they did not met all inclusion criteria (most common reason was that their neck pain could not be diagnosed as a common non specific neck pain).
Groups:
- Control: control group with no treatment only regular assessment appointments
- Spinal Manipulation: spinal manipulation
- Spinal Manipulation and Exercises: Spinal manipulation + exercises
Period: Overall Study
Arm/Group | Control | Spinal Manipulation | Spinal Manipulation and Exercises
Started | 29 | 36 | 33
Completed | 27 | 32 | 32
Not Completed | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Spinal Manipulation | Spinal Manipulation and Exercises | Total
Number analyzed (Participants) | 29 | 36 | 33 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 36 | 33 | 98
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 37 (11) | 37 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 14 | 51
  Male | 6 | 22 | 19 | 47
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 36 | 33 | 98

OUTCOME MEASURES:

1. Secondary Outcome: Fear Avoidance Belief, Quality of Life, Range of Motion
Time Frame: One year
Reporting Status: Not Posted

2. Primary Outcome: Neck Pain
Description: Visual analog pain scale (score 0-10 cm; 0 being no neck pain and 10 extreme neck pain)
Time Frame: Up to 10 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Spinal Manipulation | Spinal Manipulation and Exercises
Number analyzed (Participants) | 29 | 36 | 33
cm | 3.8 (1.9) | 3.3 (1.7) | 3.4 (1.7)

ADVERSE EVENTS:
Arm/Group | Control | Spinal Manipulation | Spinal Manipulation and Exercises
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 0/29 | 0/36 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No